CLINICAL TRIAL: NCT05906641
Title: Modulation of Secondary Bile Acids Through the Intestinal Microbiota After Consumption of a High-protein Diet.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Armando Tovar, Head of department of nutrition physiology, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 4532
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-protein diet (Experimental): Participants will receive an isocaloric diet with a distribution of 50% carbohydrates, 30% fat and 20% protein for the two-week intervention. Additionally, they will receive a dietary supplement for the second week that will contribute another 10% of protein, obtaining 30% of protein consumption in the second week.
  Interventions: Dietary Supplement: High-protein diet

INTERVENTIONS:
Dietary Supplement: High-protein diet — Protein intake will be increased to be 30% calories from protein with calcium caseinate.

SUMMARY:
This study will investigate whether changes in the gut microbiota generated after the consumption of a high protein diet in healthy subjects, modify the production of secondary bile acids. In addition, it will be seen whether a high protein intake modifies postprandial glucose response and its relationship with gut microbiota composition.

DETAILED DESCRIPTION:
The gut microbiota is a set of microorganisms that inhabit the human digestive tract and are fundamental for the health of the host. Among the functions of the gut microbiota is the production of metabolites, such as the production of secondary bile acids from primary bile acids. On the other hand, evidence has shown that the amount of protein intake can modify the composition of the gut microbiota and in turn it increase the concentration of secondary biles acids in animal models. In addition, the consumption of a high-protein diet has been related to a decrease in postprandial glucose concentrations. Therefore, the aim of this study is to evaluate changes in secondary bile acids concentration derived from gut microbiota after the consumption of a high-protein diet in healthy subjects. Subjects with a BMI between 18.5 and 24.9 kg/m2 will be selected and will be continuously monitored with a continuous glucose monitor through 15 days. During the first 7 days participants will follow an isocaloric diet (50% carbohydrates, 30% fat and 20% protein), while during the last 7 days participants will receive an intervention with a supplement of protein (calcium caseinate) which will increase their protein intake to 30% of the total energy requirement. At the initial and final visit, blood samples will be taken for determination of biochemical parameters, amino acids and primary bile acids and a stool sample will be requested for sequencing gut microbiota and determined secondary bile acids.

ELIGIBILITY:
Inclusion Criteria:

* Male and female.
* Between 18 and older
* BMI ≥ 18.5 and ≤ 24.9 kg/m2.
* Healthy
* Willing and able to sign written informed consent prior to trial entry

Exclusion Criteria:

* Have previously diagnosed with any chronic disease
* Patients with high blood pressure.
* Patients who have suffered a cardiovascular event.
* Patients with gastrointestinal diseases.
* Weight loss > 3 kg in the last 3 months.
* Catabolic diseases such as cancer and acquired immunodeficiency syndrome.
* Pregnancy status.
* Antibiotic consumption 3 months prior to the study.
* Be an undergraduate or graduate student within the Institute.
* Subjects with creatinine > 1.3 mg/dL for men and >1 mg/dL for women and ureic nitrogen > 20 mg/dL.
* Positive smoking.
* Drug treatment:

  1. Antihypertensive drugs or treatment
  2. Treatment with hypoglycemic agents or insulin and antidiabetic drugs.
  3. Treatment with statins, fibrates or other drugs to control dyslipidemia.
  4. Use of antibiotics in the three months prior to the study.
  5. Use of steroid drugs, chemotherapy, immunosuppressants, or radiation therapy.
  6. Anorexigenic or that accelerate weight loss such as sibutramine or orlistat.
  7. Probiotic, prebiotic or symbiotic supplements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in faecal microbiota composition in response to high-protein diet | baseline, 7 days and 14 days
  Changes to the faecal microbiota will be assessed on a high-protein diet compared to an isocaloric diet in a short period of time. Bacterial composition was measured by 16 ribosomal sequencing at baseline at day 7 and at the end of the second week. The relative change of each bacterial taxon was calculated based on the abundance of the given bacteria at baseline, at 7 days and after 14 days
Increase of secondary bile acids production | baseline, 7 days and 14 days
  Increase in the concentrations of lithocholic acid and deoxycholic acid in feces (mg/g of feces) measured by the method gas chromatography represented with the units micromol.

SECONDARY OUTCOMES:
Regulation of postprandial glucose response | 14 days
  Change in interstitial glucose determined by a continuous glucose monitor (mg/dL) within two weeks.
Increase in serum glucagon concentration | Baseline, 7 days and 14 days
  Change in serum glucagon concentration determined by ELISA (pg/mL)
Decrease in serum insulin concentration | Baseline, 7 days and 14 days
  Change in serum insulin concentration determined by ELISA (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Maria del Rocio Guizar-Heredia, Master, Study Chair — Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubiran; Armando R Tovar, Doctor, Principal Investigator — Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubiran; Martha Guevara-Cruz, Doctor, Study Director — Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubiran, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Aguiar Vallim TQ, Tarling EJ, Edwards PA. Pleiotropic roles of bile acids in metabolism. Cell Metab. 2013 May 7;17(5):657-69. doi: 10.1016/j.cmet.2013.03.013. Epub 2013 Apr 18. PMID 23602448
- [Result] Guzior DV, Quinn RA. Review: microbial transformations of human bile acids. Microbiome. 2021 Jun 14;9(1):140. doi: 10.1186/s40168-021-01101-1. PMID 34127070
- [Result] Zhao X, Yang X, Hang HC. Chemoproteomic Analysis of Microbiota Metabolite-Protein Targets and Mechanisms. Biochemistry. 2022 Dec 20;61(24):2822-2834. doi: 10.1021/acs.biochem.1c00758. Epub 2022 Jan 6. PMID 34989554
- [Result] Pak HH, Cummings NE, Green CL, Brinkman JA, Yu D, Tomasiewicz JL, Yang SE, Boyle C, Konon EN, Ong IM, Lamming DW. The Metabolic Response to a Low Amino Acid Diet is Independent of Diet-Induced Shifts in the Composition of the Gut Microbiome. Sci Rep. 2019 Jan 11;9(1):67. doi: 10.1038/s41598-018-37177-3. PMID 30635612
- [Result] Tirosh A, Calay ES, Tuncman G, Claiborn KC, Inouye KE, Eguchi K, Alcala M, Rathaus M, Hollander KS, Ron I, Livne R, Heianza Y, Qi L, Shai I, Garg R, Hotamisligil GS. The short-chain fatty acid propionate increases glucagon and FABP4 production, impairing insulin action in mice and humans. Sci Transl Med. 2019 Apr 24;11(489):eaav0120. doi: 10.1126/scitranslmed.aav0120. PMID 31019023
- [Result] Kumar DP, Asgharpour A, Mirshahi F, Park SH, Liu S, Imai Y, Nadler JL, Grider JR, Murthy KS, Sanyal AJ. Activation of Transmembrane Bile Acid Receptor TGR5 Modulates Pancreatic Islet alpha Cells to Promote Glucose Homeostasis. J Biol Chem. 2016 Mar 25;291(13):6626-40. doi: 10.1074/jbc.M115.699504. Epub 2016 Jan 12. PMID 26757816
- [Result] Murphy EA, Velazquez KT, Herbert KM. Influence of high-fat diet on gut microbiota: a driving force for chronic disease risk. Curr Opin Clin Nutr Metab Care. 2015 Sep;18(5):515-20. doi: 10.1097/MCO.0000000000000209. PMID 26154278
- [Result] Singh RK, Chang HW, Yan D, Lee KM, Ucmak D, Wong K, Abrouk M, Farahnik B, Nakamura M, Zhu TH, Bhutani T, Liao W. Influence of diet on the gut microbiome and implications for human health. J Transl Med. 2017 Apr 8;15(1):73. doi: 10.1186/s12967-017-1175-y. PMID 28388917
- [Result] Wei M, Huang F, Zhao L, Zhang Y, Yang W, Wang S, Li M, Han X, Ge K, Qu C, Rajani C, Xie G, Zheng X, Zhao A, Bian Z, Jia W. A dysregulated bile acid-gut microbiota axis contributes to obesity susceptibility. EBioMedicine. 2020 May;55:102766. doi: 10.1016/j.ebiom.2020.102766. Epub 2020 May 11. PMID 32408110
- [Result] Wu S, Bhat ZF, Gounder RS, Mohamed Ahmed IA, Al-Juhaimi FY, Ding Y, Bekhit AEA. Effect of Dietary Protein and Processing on Gut Microbiota-A Systematic Review. Nutrients. 2022 Jan 20;14(3):453. doi: 10.3390/nu14030453. PMID 35276812
- [Result] FOLCH J, LEES M, SLOANE STANLEY GH. A simple method for the isolation and purification of total lipides from animal tissues. J Biol Chem. 1957 May;226(1):497-509. No abstract available. PMID 13428781
- [Result] Keller S, Jahreis G. Determination of underivatised sterols and bile acid trimethyl silyl ether methyl esters by gas chromatography-mass spectrometry-single ion monitoring in faeces. J Chromatogr B Analyt Technol Biomed Life Sci. 2004 Dec 25;813(1-2):199-207. doi: 10.1016/j.jchromb.2004.09.046. PMID 15556534
- [Result] Van Elswyk ME, Weatherford CA, McNeill SH. A Systematic Review of Renal Health in Healthy Individuals Associated with Protein Intake above the US Recommended Daily Allowance in Randomized Controlled Trials and Observational Studies. Adv Nutr. 2018 Jul 1;9(4):404-418. doi: 10.1093/advances/nmy026. PMID 30032227